CLINICAL TRIAL: NCT05163769
Title: The Efficacy of a Novel Multimodal Personalized Physical and Cognitive Training System for Neurocognitive Protection and Enhancement in Older Adults
Brief Title: Physical and Cognitive Training System for Neurocognitive Protection and Enhancement in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Nanyang Technological University (Other); Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Lee Tih Shih, Associate Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021-591
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Cognitive Decline
Keywords: Cognitive Decline; Cognitive Training; Physical Training; Exergaming; Personalized; Older Adults
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multimodal Training (Experimental): The participants in the Multimodal training arm (mBCI) will undergo 48 physical and cognitive training sessions over 24 weeks on the NeeuroCycle BCI Physical and Cognitive training system. Sessions are scheduled three times a week for the first 12 weeks and then once a week for the subsequent 12 weeks. Sessions are spaced at least one day apart and will take about one hour per session.The mBCI training program will deliver cognitive training modules in tandem with a stationary cycling regime. The cognitive training program consists of six different gamified tasks that target attention, immediate/working and delayed memory, decision-making, and visuospatial abilities delivered on an electronic tablet. The cycling regime is divided into seven non-consecutive sections. The participant will be tasked to complete a cognitive training activity that will last about 2-3 minutes between each cycling session.
  Interventions: Device: NeeuroCycle Physical and Cognitive Training System
- Neurocognitive-Training only (Experimental): The participants in the Neurocognitive training-only arm (nBCI) will undergo 48 cognitive training sessions over 24 weeks on the NeeuroCycle BCI Cognitive training system. The sessions are scheduled three times a week for the first 12 weeks and then once a week for the subsequent 12 weeks. Sessions are spaced at least one day apart and will take about one hour per session. The nBCI training protocol will deliver cognitive training modules that consists of six different gamified tasks that target attention, immediate/working and delayed memory, decision-making, and visuospatial abilities delivered on an electronic tablet. Participants will navigate the virtual space of the cognitive training program by using arrow keys on the tablet.
  Interventions: Device: NeeuroCycle Cognitive Training System
- Active Control (No Intervention): The participants in the Active Control arm (AC) will undergo 48 sessions over 24 weeks. The sessions are scheduled three times a week for the first 12 weeks and then once a week for the subsequent 12 weeks. Sessions are spaced at least one day apart and will take about one hour per session. Participants in this arm will view informative documentaries on an electronic tablet and answer three general questions about documentary.

INTERVENTIONS:
Device: NeeuroCycle Physical and Cognitive Training System — The NeeuroCycle Physical and Cognitive Training System is a novel multimodal electroencephalogram (EEG)-based physical and cognitive training device. The system mainly comprises of a recumbent bicycle device and a customized four frontal electrode EEG-headband paired with the gamified NeeuroCycle cognitive training program delivered via an electronic application (app) on a tablet. The cognitive training program is built upon patented EEG-based attention, learning, and memory algorithms.
  Arms: Multimodal Training
Device: NeeuroCycle Cognitive Training System — The NeeuroCycle Cognitive Training System is a novel electroencephalogram (EEG)-based cognitive training device. The system mainly comprises of a customized four frontal electrode EEG-headband paired with the gamified NeeuroCycle cognitive training program delivered via an electronic application (app) on a tablet. The cognitive training program is built upon patented EEG-based attention, learning, and memory algorithms.
  Arms: Neurocognitive-Training only

SUMMARY:
Neurocognitive decline is a health issue that is associated with ageing. It is often irreversible from the onset. The concomitant costs of neurocognitive decline could be potentially exponential if left unchecked. Therefore, there is a need to be able to delay the onset of age-related neurocognitive decline or possibly avoid it altogether. Previous studies have shown that there is a strong positive relationship between the fitness of neurocognitive function and cognitive training. More interestingly, recent studies also suggest that combining cognitive training with physical activity may result in a better outcome for neurocognitive function as compared to only cognitive training. Anchoring on the findings of those studies, the investigators aim to develop and evaluate the efficacy of a novel personalized multimodal brain computer interface (BCI) cognitive and physical training system for neurocognitive protection and enhancement in older adults. The current study employs a three-arm randomized-controlled trial approach. The investigators hypothesize that participants in the multimodal cognitive and physical training (mBCI) group will perform significantly better than the cognitive training-only BCI (nBCI) and active control (AC) groups on the Repeated Battery for the Assessment of Neuropsychological Status (RBANS) after an initial high-intensity 36 training session period from pre- to 12 weeks post-intervention. The investigators also hypothesize that the mBCI group will perform significantly better on the RBANS than nBCI or AC groups after the consecutive high- and low-intensity periods from pre- to 24-weeks post-intervention.

DETAILED DESCRIPTION:
Neurocognitive decline is a health problem that is associated with ageing. More often than not, age-related cognitive decline may be indicative of the onset of mild cognitive impairment (MCI), or even more severe neurocognitive disorders such as Alzheimer's and Parkinson's disease-both of which will eventually lead to dementia. Cognitive decline and neurocognitive disorders can often lead to the gross deterioration in one's quality of life. Depending on the severity and duration of the onset of the neurocognitive decline, patients may experience anything from forgetfulness or learning difficulties, to major issues such as a decreased capacity for decision-making, confusion, disorientation, communication problems, and social behavioral issues. All of these issues could impede one's ability to care for one's self, which may also lead to the increased reliance and burden on caretakers.

On a global scale, it is estimated that about 46.8 million people suffer from dementia or other dementia subtypes. That number is expected to increase by 68% over the next 30 years. The current economic burden of dementia and other dementia subtypes is evaluated at $818 billion, with projections expecting cost to rise to $2 trillion by the year 2030. In Singapore specifically, the estimated cost of dementia was reported at $1.4 billion per year, with costs expecting to rise in tandem with Singapore's rapidly aging population. Given the impact and impending threats of neurocognitive decline, it is clear that intentional efforts to combat neurocognitive decline is necessary.

To date, experts in the field have yet to identify specific causes of neurocognitive decline. This is due to the heterogeneity of neurocognitive decline and the diseases associated with it. As such, it has been challenging to find definitive causes and cures for neurocognitive decline. That said, there are several risk factors associated with neurocognitive decline and dementia. Risk factors such as age and genetics are fairly predictive of neurocognitive decline, but are, by nature, unmodifiable. However, risk factors such as, but not limited to, cardiovascular problems, physical activity, cognitive training, and social engagement are possible and much easier to modify. Hence, there has been a preponderance of interventions in the field that targets those specific modifiable risk factors with the intention of manipulating current or future neurocognitive outcomes. For example, cognitive training (CT) has been a target for interventions that promote the delay and/or prevention of neurocognitive decline. Over the past few decades, CT programs in the field have evolved to computerized, gamified, and self-manned versions that usually target specific areas of cognition such as memory, attention, decision-making, inhibition, or a combination of those areas.

Similarly, physical activity (PA) has also been a target for interventions that promote the delay and/or prevention of neurocognitive decline. Studies with PA-specific interventions have also shown to positively influence neurocognitive function in patients with mild cognitive impairment, as well as those who are at risk of developing Alzheimer's Disease. Evidence also show that PA can delay the effects of neurocognitive decline in patients with existing cognitive decline, dementia, and other dementia subtypes.

Interestingly, there has been a recent surge of interventions in the field that amalgamates both PA and CT elements. This shift in direction in the field acknowledges the symbiotic relationship between CT and PA with regards to neurocognitive outcome. Many of these studies set out to investigate the effects of 'exergaming' (a portmanteau of exercise and gaming) on neurocognitive function in the older adult population with varying neurocognitive capacity ranging from healthy to declining. Exergaming interventions have shown to improve the subjects' executive function and cognitive performance after the intervention period as compared to the subject controls. The effects of exergaming interventions were also able to delay the onset of mild cognitive impairment in healthy subjects as compared to the healthy controls in some studies. That said, such programs are still limited by factors such as poor personalization capabilities, substandard controls, and high attrition rates (lack of participant engagement). Additionally, studies of such nature are far and few between in Asia, making it unclear if similar results can be replicated in an Asian-majority demographic like Singapore.

To address these issues, the current study aims to use a novel personalized multimodal physical and cognitive brain computer interface (BCI) training system to delay and/or prevent neurocognitive decline, and enhance neurocognitive function. The investigators' proposed training system integrates a stationary cycling intervention and a corresponding personalized BCI cognitive training program. The BCI cognitive training program uses machine learning technologies and elderly-friendly user-interface/user-experience (UI/UX) game design to actively track individual neurocognitive status, provide feedback in real-time, and encourage older adults to persist in training for the long term. The investigators also seek to customize the program's UI/UX by employing locally-relevant materials to reduce accessibility barriers and increase participant engagement. For the purposes of this study, all instructions and interventions will be delivered in English. However, there are plans for future iterations of this program to include other local languages to facilitate the use of the program by non-English speaking Singaporean elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Physically healthy adults from 50 to 75 years old.
2. Mini-mental state examination (MMSE) >= 24.
3. Able to travel to study site independently.
4. Literate in English.
5. BMI within acceptable range (BMI scores from 18.5 to 24.9).
6. Able to cycle on the NeeuroCycle recumbent bicycle device at a comfortable pace for a continuous period of three minutes without experiencing symptoms of severe breathlessness, fatigue, and pain.
7. Fully vaccinated against COVID-19 (Government Approved Vaccines ONLY; at least two weeks from the date of the second vaccination)

Exclusion Criteria:

1. Any known neuropsychiatric disorders (such as dementia, epilepsy or mental retardation).
2. Presence of end stage lung, cardiac, liver, and/or renal disease.
3. Experienced any cerebrovascular and/or cardiac events in the last 6 months.
4. Have active arthritis.
5. Uncorrected gross hearing, visual and/or speech impairments.
6. Prone to vertigo, motion sickness, and/or migraine episodes.
7. Highly physically active.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Repeatable Battery for the Assessement Neuropsychological Status (RBANS) | Comparison in the change of RBANS total score from pre-treatment (Week 1; Session 1) to mid-treatment (Week 12; Session 36) to post-treatment (Week 24; Session 48) among all three study arms.
  The RBANS test provides reliable and well-validated assessments of five different cognitive domains including: language, attention, visuospatial awareness, immediate, and delayed memory.

SECONDARY OUTCOMES:
Number of Adverse Events/Serious Adverse Events Reported | Throughout the intervention period (Up to 24 weeks) for all three study arms.
  To record the number of adverse events/serious adverse events reported.
Systems Usability Scale | Two intervention groups(mBCI and nBCI): Post-intervention(Week 24; Session 48)
  Participants will rate their agreeableness on 10 statements regarding their satisfaction and ease of use of the training components on a 5-point Likert scale. Participants will also answer three qualitative questions regarding their satisfaction and ease of use.

CONTACTS AND LOCATIONS:
Overall Officials: Tih Shih Lee, MD/PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Graduate Medical School, Singapore, Singapore